CLINICAL TRIAL: NCT04100863
Title: A Non-Interventional Pilot Study to Explore the Role of Gut Flora in Autism
Status: Withdrawn | Type: Observational
Why Stopped: Company focus shifted
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-006
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Autism; Autism Spectrum Disorder; Autistic Disorder; Autism, Akinetic; Autism; Atypical; Autism; Psychopathy; Autism Fragile Syndrome X; Autism With High Cognitive Abilities; Autism-Related Speech Delay; Autism, Susceptibility to, 6; Autism Spectrum Disorder High-Functioning; Autistic Thinking; Autism, Susceptibility to, X-Linked 6; Autistic Behavior
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Akinetic Mutism; Antisocial Personality Disorder; Fragile X Syndrome; Child Development Disorders, Pervasive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals with Autism: Individuals who have been diagnosed with autism
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention for this study.

SUMMARY:
This study seeks to correlate microbiome sequencing data with information provided by patients and their medical records regarding autism.

DETAILED DESCRIPTION:
The goal of this Research Study is to better understand how the genetic information in subject's microbiome correlates to the information provided in surveys and in medical records regarding autism.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by parent or legally authorized representative
2. Male or female patients age 6 and older.
3. Diagnosis of autism per DSM-V criteria (See appendix)

Exclusion Criteria:

1. Refusal by parent or legally authorized representative to sign informed consent form
2. Treatment with antibiotics within 2 weeks prior to screening
3. Treatment with probiotics within 6 weeks prior to screening
4. History of bariatric surgery, total colectomy with ileorectal anastomosis or proctocolectomy.
5. Postoperative stoma, ostomy, or ileoanal pouch
6. Participation in any experimental drug protocol within the past 12 weeks
7. Treatment with total parenteral nutrition
8. Any clinically significant evidence of disease that could interfere with the subject's ability to enter the trial
9. Inability of parent or legally authorized representative to adequately communicate with the investigator or their respective designee and/or comply with the requirements of the entire study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals ages 6 and older who have been diagnosed with Autism
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Correlation of Microbiome to Autism via Relative Abundance Found in Microbiome Sequencing | 1 year
  Relative abundance of bacterial classes within taxonomic phyla and, more broadly, within their domain will be analyzed by sequencing the gut microbiome. These data will then be categorized among specific Autism Spectrum Disorders

SECONDARY OUTCOMES:
Validation of Sequencing Methods | 1 year
  To validate the methods used to sequence samples

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only aggregated and deidentified data will be shared with other researchers.